CLINICAL TRIAL: NCT03009877
Title: Preoxygenation With Optiflow™, a High Flow Nasal Cannula (HFNC), is Superior to Preoxygenation With Facemask in Morbidly Obese Patients Undergoing General Anesthesia
Brief Title: Preoxygenation With Optiflow™ in Morbidly Obese Patients is Superior to Face Mask
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: withdrawn prior to IRB approval
Sponsor: Montefiore Medical Center (Other)
Collaborators: The University of Texas Health Science Center, Houston (Other); M.D. Anderson Cancer Center (Other)
Responsible Party: Principal Investigator, Tracey Straker, Co-principal investigator, Attending Anesthesiologist, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-7360
Record Dates: First submitted 2016-12-21; First posted 2017-01-04 (Estimated); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Obesity, Morbid
MeSH Terms: conditions — Obesity, Morbid | interventions — Masks; Rocuronium; Propofol; Fentanyl; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Preoxygenation with face mask (Active Comparator): Standard preoxygenation with a mask will be performed for five minutes. Once preoxygenation is complete, patients will be induced with standard induction medications including lidocaine, midazolam, fentanyl and propofol. Once the patient is apneic, one breath will be given via facemask to confirm ventilation and then 0.6 mg/kg of rocuronium will be administered. The 5.5mm flexible intubation scope will be introduced into the oropharynx and advanced into the trachea with the assistance of the C-MAC video laryngoscope. Once the flexible intubation scope is in the trachea, the endotracheal tube (7.0 mm unless otherwise specified) will be advanced. Ventilation will not begin until the primary or secondary endpoints are reached.
  Interventions: Device: facemask; Drug: Rocuronium; Drug: Propofol; Drug: Fentanyl; Drug: Midazolam; Device: C-MAC Premium Video Intubation Platform-KARL STORZ
- Preoxygenation via hi flow nasal cannula (Experimental): The high flow nasal cannula (Optiflow) will be applied as soon as the patient is in the operating room. The patient will be preoxygenated with high flow nasal cannula at 50 L/min for 5 minutes. After induction, general anesthesia will be maintained with a propofol infusion. One breath will be given via facemask to confirm ventilation and then 0.6 mg/kg of rocuronium will be administered. Upon apnea, the Optiflow™ flow will be increased to 70 L/min and jaw thrust will be performed until the patient is adequately relaxed. The video laryngoscope (C-MAC) will then be introduced into the oropharynx and the flexible intubation scope advanced into the trachea with the assistance of the C-MAC. Once the flexible intubation scope is in the trachea, the endotracheal tube will be advanced.
  Interventions: Device: Optiflow F&P 850™ System; Drug: Rocuronium; Drug: Propofol; Drug: Fentanyl; Drug: Midazolam; Device: C-MAC Premium Video Intubation Platform-KARL STORZ

INTERVENTIONS:
Device: Optiflow F&P 850™ System — Optiflow™ (Fisher & Paykel Healthcare Limited, East Tamaki, Auckland-New Zealand) offers the ability to comfortably deliver a complete range of oxygen concentrations and flows to extend the traditional boundaries of oxygen therapy.
  This will be placed on the patient immediately upon entering the operating room for 5 minutes, at 50 liters per minute then increased to 70 liters per minute after induction.
  Other Names: High flow nasal cannula
  Arms: Preoxygenation via hi flow nasal cannula
Device: facemask — We will apply the facemask to the patient immediately upon entering the operating room to pre-oxygenate for five minutes.
  Other Names: face mask
  Arms: Preoxygenation with face mask
Drug: Rocuronium — Rocuronium will be administered after the ability to mask ventilate is determined.
Drug: Propofol — Propofol infusion 50 micrograms to 150 micrograms will be administered immediately on induction to maintain sedation throughout apneic oxygenation.
Drug: Fentanyl — Fentanyl will be administered at the beginning of induction, 2 micrograms per kilogram.
Drug: Midazolam — midazolam will be given upon induction, 1-2 milligrams at the anesthesiologist's discretion.
  Other Names: Versed
Device: C-MAC Premium Video Intubation Platform-KARL STORZ — After patient is induced, the 5.5mm flexible intubation video scope (C-MAC Premium Video Intubation Platform-KARL STORZ) will then be introduced into the oropharynx and advanced into the trachea with the assistance of the C-MAC video laryngoscope (3 or 4 blade based on anesthesiologist's discretion).
  Other Names: videolaryngoscope and optical fiberoptic bronchoscope

SUMMARY:
Optiflow™ may provide an opportunity to prolong apnea time in the morbidly obese patient population. This study will examine whether Optiflow can do this, and compare the pre-oxygenation with Optiflow to the pre-oxygenation achieved with face mask.

DETAILED DESCRIPTION:
The use of high flow nasal cannula (HFNC) originated in neonatal care, and has become widespread in its application for patients that are high risk for hypoxemia, both in critical care and emergency settings. Therefore, high flow nasal oxygenation continues to be studied in airway management for preoxygenation, as well as maintenance of oxygenation in airway procedures. Optiflow™, a humidified high flow nasal cannula, has already been shown to be useful in preventing desaturation during intubation in ICU patients versus the non-rebreathing mask, in addition to, prolonging safe apnea time in patients with potential difficult airways. Additionally, preoxygenation with HFNC prior to intubation of patients in hypoxemic respiratory failure has also been shown to decrease desaturation during apnea compared to preoxygenation with traditional bag valve mask. The morbidly obese patient presents a separate group of challenges to the anesthesiologist in regards to mask ventilation and intubation. Obesity (along with other factors) has been shown to contribute to difficulty with mask ventilation. Obese patients have altered respiratory physiology, including decreased functional residual capacity, increased oxygen consumption and lower tidal volumes, as compared to the non-obese patient. These factors contribute to obese patients potentially having a shorter apnea time before desaturating during induction of general anesthesia, as compared to the non-obese patient. Weight is inversely correlated with safe apnea time. Optiflow™ may provide an opportunity to prolong apnea time in the morbidly obese patient population. If demonstrated to be efficacious as a method for preoxygenation and prolongation of apneic time, this could provide a safer environment for intubation in this particular patient population.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years old) undergoing elective surgery requiring general anesthesia
* BMI > 40 kg/m2
* American Society of Anesthesiology (ASA) Physical Status II-III

Exclusion Criteria:

* Chronic hypoxemia (SpO2 <94% on room air or on home oxygen)
* Acute respiratory failure
* Coronary artery disease and/or congestive heart failure
* Moderate-Severe pulmonary hypertension and/or RV dysfunction
* Full stomach (recently eaten)
* Pregnancy
* Chronic pulmonary disease (specifically COPD or interstitial disease, NOT asthma)
* Respiratory tract pathology
* Facial Abnormality
* American Society of Anesthesiology (ASA) Physical Status IV-V

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-07 (Estimated); Primary Completion 2019-05 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Time to desaturation | up to 10 minutes
  Intraoperatively, apneic time will be record from the time of administration of the muscle relaxant. The time until the first desaturation will be recorded. The maximum time of measurement will be 10 minutes.

SECONDARY OUTCOMES:
Time until hypercarbia > 65 mmHg | up to 10 minutes
  The time until hypercarbia to more than 65 mmHg will be measured from the time of administration of the muscle relaxant. The time until transcutaneous CO2 is > 65 mmHg will be recorded, unless 10 minutes is reached before that level is reached.
Assess correlation between end tidal CO2 and transcutaneous CO2 monitoring | up to 10 minutes
  Assessment of accurate correlation between transcutaneous CO2 monitoring, end tidal CO2, and/or PaCO2 will be performed up to 10 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Irene Osborn, MD, Study Director — Montefiore Medical Center

IPD SHARING:
Plan to Share IPD: Yes
This is a collaborative study, so the information will be shared with the researchers in Texas. However, we do not plan to use this information for other studies.

REFERENCES:
- [Background] Locke RG, Wolfson MR, Shaffer TH, Rubenstein SD, Greenspan JS. Inadvertent administration of positive end-distending pressure during nasal cannula flow. Pediatrics. 1993 Jan;91(1):135-8. PMID 8416477
- [Background] Frat JP, Thille AW, Mercat A, Girault C, Ragot S, Perbet S, Prat G, Boulain T, Morawiec E, Cottereau A, Devaquet J, Nseir S, Razazi K, Mira JP, Argaud L, Chakarian JC, Ricard JD, Wittebole X, Chevalier S, Herbland A, Fartoukh M, Constantin JM, Tonnelier JM, Pierrot M, Mathonnet A, Beduneau G, Deletage-Metreau C, Richard JC, Brochard L, Robert R; FLORALI Study Group; REVA Network. High-flow oxygen through nasal cannula in acute hypoxemic respiratory failure. N Engl J Med. 2015 Jun 4;372(23):2185-96. doi: 10.1056/NEJMoa1503326. Epub 2015 May 17. PMID 25981908
- [Background] Hayes-Bradley C, Lewis A, Burns B, Miller M. Efficacy of Nasal Cannula Oxygen as a Preoxygenation Adjunct in Emergency Airway Management. Ann Emerg Med. 2016 Aug;68(2):174-80. doi: 10.1016/j.annemergmed.2015.11.012. Epub 2015 Dec 31. PMID 26747218
- [Background] Badiger S, John M, Fearnley RA, Ahmad I. Optimizing oxygenation and intubation conditions during awake fibre-optic intubation using a high-flow nasal oxygen-delivery system. Br J Anaesth. 2015 Oct;115(4):629-32. doi: 10.1093/bja/aev262. Epub 2015 Aug 7. PMID 26253608
- [Background] Simon M, Braune S, Frings D, Wiontzek AK, Klose H, Kluge S. High-flow nasal cannula oxygen versus non-invasive ventilation in patients with acute hypoxaemic respiratory failure undergoing flexible bronchoscopy--a prospective randomised trial. Crit Care. 2014 Dec 22;18(6):712. doi: 10.1186/s13054-014-0712-9. PMID 25529351
- [Background] Miyagi K, Haranaga S, Higa F, Tateyama M, Fujita J. Implementation of bronchoalveolar lavage using a high-flow nasal cannula in five cases of acute respiratory failure. Respir Investig. 2014 Sep;52(5):310-4. doi: 10.1016/j.resinv.2014.06.006. Epub 2014 Jul 25. PMID 25169847
- [Background] Gottschalk A, Mirza N, Weinstein GS, Edwards MW. Capnography during jet ventilation for laryngoscopy. Anesth Analg. 1997 Jul;85(1):155-9. doi: 10.1097/00000539-199707000-00028. PMID 9212140
- [Background] Nishimura M. High-flow nasal cannula oxygen therapy in adults. J Intensive Care. 2015 Mar 31;3(1):15. doi: 10.1186/s40560-015-0084-5. eCollection 2015. PMID 25866645
- [Background] Patel A, Nouraei SA. Transnasal Humidified Rapid-Insufflation Ventilatory Exchange (THRIVE): a physiological method of increasing apnoea time in patients with difficult airways. Anaesthesia. 2015 Mar;70(3):323-9. doi: 10.1111/anae.12923. Epub 2014 Nov 10. PMID 25388828
- [Background] Maggiore SM, Idone FA, Vaschetto R, Festa R, Cataldo A, Antonicelli F, Montini L, De Gaetano A, Navalesi P, Antonelli M. Nasal high-flow versus Venturi mask oxygen therapy after extubation. Effects on oxygenation, comfort, and clinical outcome. Am J Respir Crit Care Med. 2014 Aug 1;190(3):282-8. doi: 10.1164/rccm.201402-0364OC. PMID 25003980
- [Background] Aceto P, Perilli V, Modesti C, Ciocchetti P, Vitale F, Sollazzi L. Airway management in obese patients. Surg Obes Relat Dis. 2013 Sep-Oct;9(5):809-15. doi: 10.1016/j.soard.2013.04.013. Epub 2013 May 6. PMID 23810609
- [Background] Murphy C, Wong DT. Airway management and oxygenation in obese patients. Can J Anaesth. 2013 Sep;60(9):929-45. doi: 10.1007/s12630-013-9991-x. Epub 2013 Jul 9. PMID 23836064
- [Background] Sinha A, Jayaraman L, Punhani D. ProSeal LMA increases safe apnea period in morbidly obese patients undergoing surgery under general anesthesia. Obes Surg. 2013 Apr;23(4):580-4. doi: 10.1007/s11695-012-0833-7. PMID 23361469
- [Background] Jense HG, Dubin SA, Silverstein PI, O'Leary-Escolas U. Effect of obesity on safe duration of apnea in anesthetized humans. Anesth Analg. 1991 Jan;72(1):89-93. doi: 10.1213/00000539-199101000-00016. PMID 1984382
- [Background] Gambee AM, Hertzka RE, Fisher DM. Preoxygenation techniques: comparison of three minutes and four breaths. Anesth Analg. 1987 May;66(5):468-70. No abstract available. PMID 3578856
- [Background] Tang L, Li S, Huang S, Ma H, Wang Z. Desaturation following rapid sequence induction using succinylcholine vs. rocuronium in overweight patients. Acta Anaesthesiol Scand. 2011 Feb;55(2):203-8. doi: 10.1111/j.1399-6576.2010.02365.x. PMID 21226862
- [Background] Dixon BJ, Dixon JB, Carden JR, Burn AJ, Schachter LM, Playfair JM, Laurie CP, O'Brien PE. Preoxygenation is more effective in the 25 degrees head-up position than in the supine position in severely obese patients: a randomized controlled study. Anesthesiology. 2005 Jun;102(6):1110-5; discussion 5A. doi: 10.1097/00000542-200506000-00009. PMID 15915022
- [Background] Boyce JR, Ness T, Castroman P, Gleysteen JJ. A preliminary study of the optimal anesthesia positioning for the morbidly obese patient. Obes Surg. 2003 Feb;13(1):4-9. doi: 10.1381/096089203321136511. PMID 12630606
- [Background] Simon M, Wachs C, Braune S, de Heer G, Frings D, Kluge S. High-Flow Nasal Cannula Versus Bag-Valve-Mask for Preoxygenation Before Intubation in Subjects With Hypoxemic Respiratory Failure. Respir Care. 2016 Sep;61(9):1160-7. doi: 10.4187/respcare.04413. Epub 2016 Jun 7. PMID 27274092
- [Background] Teller LE, Alexander CM, Frumin MJ, Gross JB. Pharyngeal insufflation of oxygen prevents arterial desaturation during apnea. Anesthesiology. 1988 Dec;69(6):980-2. doi: 10.1097/00000542-198812000-00035. No abstract available. PMID 3195773
- [Background] Taha SK, Siddik-Sayyid SM, El-Khatib MF, Dagher CM, Hakki MA, Baraka AS. Nasopharyngeal oxygen insufflation following pre-oxygenation using the four deep breath technique. Anaesthesia. 2006 May;61(5):427-30. doi: 10.1111/j.1365-2044.2006.04610.x. PMID 16674614
- [Background] Ramachandran SK, Cosnowski A, Shanks A, Turner CR. Apneic oxygenation during prolonged laryngoscopy in obese patients: a randomized, controlled trial of nasal oxygen administration. J Clin Anesth. 2010 May;22(3):164-8. doi: 10.1016/j.jclinane.2009.05.006. PMID 20400000